CLINICAL TRIAL: NCT03008382
Title: Interstitial Cystitis: Examination of the Central Autonomic Network
Acronym: ICECAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Endeavor Health (Other); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Thomas Chelimsky, MD, Director, VCU Comprehensive Autonomic Center; Director, 4PCP Curriculum (Primary Practice Practitioner Program for Chronic Pain), Virginia Commonwealth University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HM20025835
Record Dates: First submitted 2016-12-28; First posted 2017-01-02 (Estimated); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Interstitial Cystitis/Painful Bladder Syndrome; Myofascial Pelvic Pain
Keywords: Interstitial Cystitis; Pelvic Pain
MeSH Terms: conditions — Cystitis, Interstitial; Pelvic Pain | interventions — Metoprolol

STUDY DESIGN:
Intervention Model Description: Participants with Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS) and/or Myofascial Pelvic Pain (MPP) will be randomized to take 8 weeks of Metoprolol Tartrate Oral Tablet or Placebo Oral Tablet, followed by a 4-Week washout period, and then 8 weeks of Placebo or Metoprolol.
Who Masked: Participant, Investigator
Masking Description: Participants and investigator did not know if they were randomized to intervention or placebo first for Chronic pelvic pain group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Chronic Pelvic Pain (Other): Participants with chronic pelvic pain will be randomized to either take 8 weeks of Metoprolol Tartrate Oral Tablet, followed by a 4-Week washout period, and then 8 weeks of Placebo OR to take 8 weeks of Placebo Oral Tablet, followed by a 4-Week washout period, and then 8 weeks of Metoprolol Tartrate Oral Tablet. This intervention aims at determining whether Metoprolol reduces pain in subjects in both groups compared to placebo. Some participants were not randomized and were instead enrolled into the observational sub-study.
  Interventions: Drug: Metoprolol Tartrate Oral Tablet; Drug: Placebo Oral Tablet; Other: No intervention- observational sub-study
- Healthy Control Group (No Intervention): Healthy female subjects ages 18-80 with various demographic background who do not have any exclusionary diagnostic or symptomatic criteria will be recruited. Subjects will never receive any randomization or drug treatment during the entire duration of the study

INTERVENTIONS:
Drug: Metoprolol Tartrate Oral Tablet — Metoprolol is a beta-blocker commonly used for mild blood pressure control, and also commonly used for migraine. Subjects with IC/BPS or MPP will start metoprolol at 25 mg once daily and increase to the goal dose of 25 mg 2/day after one week and continue for 8 weeks total.
  Other Names: Metoprolol
  Arms: Chronic Pelvic Pain
Drug: Placebo Oral Tablet — Subjects with IC/BPS or MPP will start placebo distributed in a double-blind manner. Subjects will take placebo once daily and increase to the goal dose of 25 mg 2/day after one week and continue for 8 weeks total.
  Other Names: Placebo
  Arms: Chronic Pelvic Pain
Other: No intervention- observational sub-study — Participants did not receive placebo or metoprolol during the entire duration of the study.
  Arms: Chronic Pelvic Pain

SUMMARY:
This proposal aims to move the science of chronic pelvic pain (CPP) from simple associations towards an investigation of cause and effect relationships. The investigators will determine whether the striking changes in autonomic nervous system responsiveness (ANS-R) contribute meaningfully to the pathogenesis of CPP.

DETAILED DESCRIPTION:
This multi-site trial will recruit 2 groups of female subjects ages 18-80 years, evenly distributed across decades (10 or 20 per decade as appropriate): Chronic pelvic pain (CPP) and Healthy Controls (HC). The chronic pelvic pain group will be split into 2 sub groups where some participants will receive metopropol then placebo while the other participants in this interventional group will receive placebo then metoprolol.

This proposal aims to move the science of chronic pelvic pain (CPP) from simple associations towards an investigation of cause and effect relationships. We will determine whether the striking changes in ANS-R contribute meaningfully to the pathogenesis of CPP through 3 aims:

1. Careful longitudinal repeated measures in individual subjects to determine if ANS-R changes precede clinical changes;
2. Assessing the impact of an intervention designed to change ANS-R on the clinical course of CPP;
3. Evaluating changes in brain connectivity between the prefrontal cortex (PFC) and the periaqueductal gray (PAG) associated with changes in ANS-R and improved disease status.

Subjects will be pre-screened in person or on the phone. An in-person pre-screen takes place in the MCW Neurology Research Rooms at Froedtert Hospital. If the subject is able to participate, subject will sign the informed consent form before completing a baseline evaluation. The baseline evaluation occurs either following consent or at another date convenient for them. Subjects must complete all baseline activities within 2 weeks, or before their Week 4/Visit 2. The baseline evaluation is comprised of a general examination, a set of questionnaires, background history documenting date of diagnosis, medications tried, duration of each treatment and dosing, surgeries and therapeutic and exploratory procedures performed. A pelvic examination will be performed with CPP subjects patients only. Active Change in Posture (ACP) is administered to the subject. Subjects will complete the uroflow (urine) measurement and Valsalva maneuver in the MCW Neurology Research Rooms with a member of the research team present.

Observational Substudy:

This substudy is identical to the above with the exception of not taking a beta-blocker or placebo and is only 12 weeks long instead of 24. This is strictly an observational study to monitor subjects who have been diagnosed with IC or MPP. If the screening information shows that the subject meets the requirements, then they will be able to start. If the screening information shows that they cannot be in the research, the research doctor will discuss other options with them and/or refer them back to their regular doctor.

If the subject is able to participate, they will complete 3 regular on-site long-visits at weeks 0, 4, and 12. The first long-visit (baseline evaluation) may occur either today following consent or at another date convenient for them. The baseline evaluation comprises a general and pelvic examination (no speculum), psychological questionnaires and a background history questionnaire.

Weekly Home Checks will occur for 24 weeks (or 12 weeks if in observational sub-study) following consent. Once each a week, subjects will complete a 24-hour heart rate (HR) recording and the ACP recording using the eMotion Faros 360° portable EKG device. A member of the research team will contact the subject each week while they complete the weekly questionnaires and ACP recording. This will ensure compliance and will give the subject the opportunity to ask any questions.The researcher will remain on the phone or via Skype to monitor the subject while the ACP recording is completed from home just prior to the subject's bedtime. The HR recording will be uploaded to MCW's secure server at the subject's next hospital visit. Throughout the study, subjects flare activity will be monitored via phone calls and recording flares in the EMA application on the smartphone. This will be a Daily Flare Question in the EMA which is a set alarmed time to sound as a reminder for the duration of the subject's participation.

The following weeks after each site visit and the night before visit 5, subjects will repeat complete the 24-hr HR recording to ensure comparability of the HRV recording at home to the one performed at the matching on-site visit., Subjects will also complete the 24-h voiding diary, a set of questions using the ICECAN mobile App installed on a pre-loaded smartphone and questionnaires. Deidentified 24-hour HRV and ACP recordings will be sent to Ohio State University for analysis.

Follow-up Visits: Weeks 4, 12, 16, 24, Visits 2-5 (weeks 4 and 12 (Visits 2 and 3) for the observational substudy) Subjects will arrive to MCW Neurology Research Rooms to repeat the following: review of comorbidities, tender points exam, questionnaires, ACP and DNIC tests. Subjects will complete the Valsalva maneuver in the MCW Neurology Research Rooms with a member of the research team present. Chronic Pelvic Pain patients subjects will complete a repeat pelvic examination at Weeks 12 and 24.

CPP aparticipants will be randomized to receive 8 weeks of either placebo (a pill with no active agent), or metoprolol (a pill that reduces the impact of the brain's "fight or flight" circuits). Metoprolol is in the class of "beta-blockers" commonly used for mild blood pressure control, and also commonly used for migraine. Subjects will be administered 8 weeks of metoprolol or placebo starting at their Week 4 Visit. Subjects will complete a 4-week washout period (Week 12-16) and will be administered 8 weeks of crossover (Weeks 16-24).

Blood will be drawn (~ 50 mL, a little more than 3 tablespoons) at each in-person visit at weeks 0, 4, 12, 16, and 24 for chronic pelvic pain subjects (healthy control only at Baseline and Final visits; 2 draws total). A portion of the blood plasma/serum will be sent to the University of Pittsburgh for additional related analysis. The sample will be labeled by a number and will not contain any information that can be used to directly identify subject. This portion of the study is critical to gather new information about pelvic pain, which is very poorly understood and we highly encourage subjects to participate in this portion of the study; however, it is optional.

Healthy Controls:

60 healthy control subjects will also complete this study in 24 weeks that include 4 long site visits and 6 weekly home check visits. During this first long visit they will complete a general exam and physician evaluation, DNIC, ACP, Valsalva maneuver, and questionnaires. Subjects will complete a 24-hour HR recording from home once a week for 6 weeks total.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 80 years old
* Healthy controls; Patients diagnosed with Interstitial cystitis/Painful bladder syndrome (IC/BPS) or Myofascial pelvic pain (MPP)
* IC/BPS - ≥3 months chronic pelvic pain, pressure or discomfort perceived to be related to the urinary bladder accompanied by at least one other urinary symptom like persistent urge to void or frequency. Confusable diseases as the cause of the symptoms must be excluded, particularly recurrent UTI
* MPP - ≥3 months of non-cyclic continuous pelvic pain unrelated to bladder state and a minimum of 2 of 5 examined pelvic floor TPs scoring at least 4 out of 10 on a numeric rating scale using 2 kg pressure applied with the index finger
* Provision of informed consent prior to any study specific procedures

Exclusion Criteria:

* Known nervous system conditions including but not limited to diabetic neuropathy, Parkinson's disease, Alzheimer's disease, multiple sclerosis, strokes, seizures, etc.
* Baseline heart rate < 50 bpm; blood pressure ≥ 140/80 mmHg at rest or uncontrolled hypertension; or hypertension requiring more than two drugs for control
* Pregnant, attempting to become pregnant , or breast-feeding
* Unevaluated hematuria or infection at the time of enrollment
* Pelvic or bladder neoplasm or infection
* Severe asthma, inflammatory arthritis, connective tissue or auto-immune disorders
* Evidence of unstable medical disorder such as kidney (rising creatinine or end-stage renal failure) or liver impairment (rising AST or ALT, or end-stage with coagulopathy); poorly controlled significant cardiovascular (CHF), respiratory, endocrine (diabetes - A1c > 9 - or untreated thyroid dysfunction) or uncontrolled psychiatric illness (such as untreated depression, psychosis, etc.)
* Treatment with a drug or medical device within the previous 30 days that has not received regulatory approval
* Use of hormones (except insulin, thyroid replacement or oral contraceptives). Hormone replacement therapy is acceptable
* Current, ongoing drug or alcohol abuse
* Current use of 150 mg or more of narcotics or morphine equivalent (or inconsistent dosages or frequency - varying by > 50 mg morphine equivalent per day)
* Previous augmentation cystoplasty, cystectomy, cytolysis, or neurectomy. Pelvic surgery in the last 6 months.
* Any major surgical intervention with general anesthesia in the last 90 days. Current use of anticholinergic medications.
* Current use of beta-blocker(s).
* Unwillingness to take a beta blocker and placebo, or planned use of beta-blocker(s) other than study medication.
* Previous allergic or serious reaction to beta-blockers. Initiation of neural stimulator in the last 30 days.
* Any on-going or pending medical, health or disability related litigation, or current pursuit of disability.
* Any condition that in the judgment of the investigator and the internal advisory panel would interfere with the patient's ability to provide informed consent, comply with study instructions, place the patient at increased risk, or which would clearly confound the interpretation of the study results (specific reason will be documented).
* Current participation in another clinical trial that interferes with ICECAN policies and procedures .
* Investigators, study staff and their immediate families.
* Inability to speak, read, and understand English.
* Allergy to adhesives.
* Initiation of any new treatment class in the last 30 days, or intent to initiate a new class of treatment in the study. Treatment classes include:

  1. Pelvic injection
  2. Pelvic floor therapy
  3. Agents with specific FDA approval for IC/BPS or MPP (e.g., Elmiron)
  4. Anticonvulsants
  5. Tricyclic agents
  6. Intravesical therapy or Botox
  7. Bladder hydrodistention

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Chelimsky, MD, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - NorthShore University HealthSystem, Evanston, Illinois
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
All participant data will be de-identified before sharing.
  Blood and Urine: A portion of the blood plasma/serum and urine will be sent to the University of Pittsburgh for additional related analysis.
  Heart Rate Variability (HRV): 24-hour HRV and Active Change of Posture recordings will be sent to Ohio State University for analysis.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The participant's collected data is de-identified immediately. The blood and urine are stored in a freezer until there are enough samples to send out for analysis.
  Heart rate recordings are uploaded to a secure MCW storage site and shared for analysis throughout the participant's participation.
Access Criteria: Participant data will be shared through a secured web dropbox called BOX. BOX access is paid for and controlled by the Medical College of Wisconsin (MCW). The folders containing participant data are password protected and only those who are adding to the folders or performing analysis on collected data are given access through MCW.
  MCW's other two recruiting sites, NorthShore University HealthSystem and Case Western Reserve University, are able to add participant data to their own site folders, and each site only has access to their participants' data.
  Ohio State University has access to the folder containing participants' heart rate recording to perform analysis.
  Blood and Urine samples are deidentified and stored at MCW until a shipment is prepared. They are then sent to the University of Pittsburgh for further analysis.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was modified to report data for participants with IC/BPS and MPP as a single combined chronic pelvic pain group. Please review the pre-assignment details sections to view how participants are being presented in for this group.
Pre-assignment Details: Participants enrolled into the Chronic Pain Group were randomized into 2 sequences or were enrolled into the observational study group: "Metopropol then Placebo," "Placebo then Metopropol OR "Observational Participants." The "participant flow" and "baseline characteristics" sections for the Chronic Pain Group are presented per sequence.
Groups:
- Metoprolol Then Placebo: Participants will be randomized to take 8 weeks of Metoprolol Tartrate Oral Tablet followed by a 4-Week washout period, and then 8 weeks of Placebo.
- Placebo Then Metoprolol: Participants will be randomized to take 8 weeks of Placebo followed by a 4-Week washout period, and then 8 weeks of Metoprolol Tartrate Oral Tablet.
- Healthy Control: Healthy female subjects ages 18-80 with various demographic background who do not have any exclusionary diagnostic or symptomatic criteria will be recruited. Subjects will never receive any randomization or drug treatment during the entire duration of the study Placebo Oral Tablet: Subjects with IC/BPS or MPP will start placebo distributed in a double-blind manner. Subjects will take placebo once daily and increase to the goal dose of 25 mg 2/day after one week and continue for 8 weeks total.
- Observational Participants: Participants who meet the study eligibility criteria but were not randomized into the two interventional sequences. Participants were not randomized and did not receive any study drugs during the entire duration of the study.
Period: Overall Study
Arm/Group | Metoprolol Then Placebo | Placebo Then Metoprolol | Healthy Control | Observational Participants
Started | 23 | 22 | 23 | 4
Completed | 20 | 16 | 18 | 4
Not Completed | 3 | 6 | 5 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrew from study but did not withdraw consent | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Screenfail | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Control: Healthy female subjects ages 18-80 with various demographic background who do not have any exclusionary diagnostic or symptomatic criteria will be recruited. Subjects will never receive any randomization or drug treatment during the entire duration of the study.
- Total: Total of all reporting groups
Arm/Group | Metoprolol Then Placebo | Placebo Then Metoprolol | Healthy Control | Observational Participants | Total
Number analyzed (Participants) | 23 | 22 | 23 | 4 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 22 | 22 | 3 | 70
  >=65 years | 0 | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 23 | 4 | 72
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 12 | 14 | 8 | 2 | 36
  Unknown or Not Reported | 10 | 7 | 15 | 2 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 0 | 4
  White | 12 | 13 | 6 | 2 | 33
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 7 | 15 | 2 | 34
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 23 | 4 | 72

OUTCOME MEASURES:

1. Primary Outcome: Total Score on Genitourinary Pain Index (GUPI) Scale
Description: The total GUPI score is calculated from the sum of the 3 scores from the subscales. There is no uniformity in the ranges of scores for the individual questions. The 3 subscales are: pain, urinary, and quality of life. The total score range can go from 0-45. The higher the score indicates more female urinary symptoms. Scores were calculated for each participant at weeks 4 (baseline), 12 (post-first intervention) and 24 (post-second intervention) of their participation in the study.
Time Frame: Weeks 4, 12 and 24
Population: This assessment was not administered to all participants at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Metoprolol Then Placebo; Placebo Then Metoprolol: Participants with Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS) and/or Myofascial Pelvic Pain (MPP) will be randomized to take 8 weeks of Metoprolol Tartrate Oral Tablet or Placebo Oral Tablet, followed by a 4-Week washout period, and then 8 weeks of Placebo or Metoprolol. This intervention aims at determining whether Metoprolol reduces pain in subjects in both groups compared to placebo.
  Metoprolol Tartrate Oral Tablet: Metoprolol is a beta-blocker commonly used for mild blood pressure control, and also commonly used for migraine. Subjects with IC/BPS or MPP will start metoprolol at 25 mg once daily and increase to the goal dose of 25 mg 2/day after one week and continue for 8 weeks total.
  Placebo Oral Tablet: Subjects with IC/BPS or MPP will start placebo distributed in a double-blind manner. Subjects will take placebo once daily and increase to the goal dose of 25 mg 2/day after one week and continue for 8 weeks total.
Arm/Group | Metoprolol Then Placebo | Placebo Then Metoprolol | Healthy Control | Observational Participants
Number analyzed (Participants) | 21 | 21 | 17 | 4
score on a scale
  Week 4 | 24.4 (8.54) | 22.2 (8.94) | 2.35 (2.37) | 29.25 (7.27)
  Week 12: number analyzed (Participants) | 20 | 18 | 8 | 4
  Week 12 | 22.8 (11.1) | 21.4 (8.88) | 2.42 (3.67) | 26.65 (9.84)
  Week 24: number analyzed (Participants) | 19 | 14 | 3 | 0
  Week 24 | 23.1 (12) | 22.1 (7.8) | 1.67 (1.15) |

2. Primary Outcome: Average Score on the First Domain of the Multidimensional Pain Scoring (MPI) Scale
Description: The average score comes from the Pain Experience, the first domain, of the MPI. Domain 1 includes five scales designed to measure important dimensions of the chronic pain experience including; 1) perceived interference of pain in vocational, social/recreational, and family/marital functioning, 2) support or concern from spouse or significant other, 3) pain severity, 4) perceived life control, and 5) affective distress. Higher scores indicate more impactful effects of the pain experience in daily life. Responses from individual questions range from 0-6. 0 indicated no pain/no interference/no change. 6 indicates very intense pain/extreme interference/extreme change. The final total score range is 0-6 with 0 being absent pain and 6 being the worst pain rating. A lower score is better. Scores were calculated for each participant at weeks 4 (baseline), 12 (post-first intervention) and 24 (post-second intervention) of their participation in the study.
Time Frame: Weeks 4, 12 and 24
Population: This assessment was not administered to all participants at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Metoprolol Then Placebo | Placebo Then Metoprolol | Healthy Control | Observational Participants
Number analyzed (Participants) | 22 | 21 | 17 | 4
score on a scale
  Week 4 | 2.44 (1.11) | 2.16 (0.878) | 1.28 (0.28) | 2.95 (1.38)
  Week 12: number analyzed (Participants) | 20 | 18 | 8 | 4
  Week 12 | 2.53 (1.03) | 1.99 (0.863) | 1.41 (0.45) | 2.57 (1.42)
  Week 24: number analyzed (Participants) | 19 | 14 | 3 | 0
  Week 24 | 2.35 (1.14) | 2.11 (0.747) | 1.13 (0.35) |

3. Other Pre Specified Outcome: Correlation Between the Change in Autonomic Nervous System Responsiveness (ANS-R) and the Change in the Connectivity Between Prefrontal Cortex (PFC) and Periaqueductal Gray (PAG)
Description: A linear model with connectivity at 24 weeks as outcome, connectivity at baseline as a covariate and change in ANS-R, demographics such as age and group and the interactions of group with other covariate.
Time Frame: 24 Weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Assessing Central Autonomic Network Connectivity in Subjects With Chronic Pelvic Pain
Description: This exploratory aim for the sub-studyused functional MRI brain imaging to examine the evolution of the connectivity of the main autonomic processing nucleus, the periaqueductal gray region, with other cortical brain regions
Time Frame: Baseline, 12 weeks and 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 weeks (duration of study)
Description: Adverse events were divided into 4 categories: Metoprolol, Placebo, Baseline Period (prior to either intervention) and Washout Period (in between the two interventions) for the randomized Chronic Pelvic Pain participants.
Groups:
- Metoprolol: Participants who experienced an adverse event while on the metoprolol intervention.
- Placebo: Participants who experienced an adverse event while on the placebo intervention.
- Baseline Period: Participants who experienced an adverse event prior to either intervention while on the study. This was during weeks 0-4 of the study.
- Washout Period: Participants who experienced an adverse event who were between interventions while on the study. This was during weeks 13-16 of the study.
- Observational Participants: Healthy female subjects ages 18-80 with various demographic background who do not have any exclusionary diagnostic or symptomatic criteria will be recruited. Subjects will never receive any randomization or drug treatment during the entire duration of the study.
- Healthy Control: Participants who meet the study eligibility criteria but were not randomized into the two interventional sequences. Participants were not randomized and did not receive any study drugs during the entire duration of the study.
Arm/Group | Metoprolol | Placebo | Baseline Period | Washout Period | Observational Participants | Healthy Control
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/42 | 0/45 | 0/40 | 0/4 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42 | 0/45 | 0/40 | 0/4 | 0/23
Other Adverse Events (participants affected / at risk) | 22/43 | 25/42 | 5/45 | 4/40 | 0/4 | 0/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metoprolol (N=43) | Placebo (N=42) | Baseline Period (N=45) | Washout Period (N=40) | Observational Participants (N=4) | Healthy Control (N=23)
Near Syncopal Event (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood post 1st round of study medication (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Yeast infection (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Worsening Bladder Pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
toothache (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep paralysis + Nightmares (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
low heart rate (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvectomy and LEEP (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reaction to lidocaine (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Car accident (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vestibular migraines with vertigo (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Valsalva maneuver-headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibromyalgia flare (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing with bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
stomach rash (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heightened mood/depressive symptoms (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder flare (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
electrode reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (allergic reaction) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hair loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
erratic sleep (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
fatigue (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats & changes in mood (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sexual dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal EKG (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lightheadedness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory issues (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wooziness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of appetite (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep problems (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
All diagnosed subjects were combined because of inadequate recruitment related to the COVID 19 pandemic which halted study recruitment. As a result, the study was no longer adequately powered to compare the differing groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT03008382/Prot_SAP_001.pdf
  • Informed Consent Form (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT03008382/ICF_000.pdf